CLINICAL TRIAL: NCT04783974
Title: Correlation Between Peri-implantitis and Assumptions of Medications: a Retrospective Study
Brief Title: Correlation Between Peri-implantitis and Assumptions of Medications
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: SC-AA-2
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-07

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients assuming SSRI: Patients treated with dental implants and assuming selective serotonin reuptake inhibitors
  Interventions: Device: Dental implants
- Patients assuming PPI: Patients treated with dental implants and assuming proton pump blockers
  Interventions: Device: Dental implants
- Patients assuming Anti-inflammatory drugs: Patients treated with dental implants and assuming anti-inflammatory drugs
  Interventions: Device: Dental implants
- Patients assuming Anti-hypertensive drugs: Patients treated with dental implants and assuming anti-hypertensive drugs
  Interventions: Device: Dental implants
- Control group - Patients not assuming the studied drugs: Patients treated with dental implants and not assuming any of the following drugs: selective serotonin reuptake inhibitors, proton pump blockers, anti-inflammatory drugs, anti-hypertensive drugs
  Interventions: Device: Dental implants

INTERVENTIONS:
Device: Dental implants — Treatment of total or partial edentulism through the placement of osseointegrated dental implants

SUMMARY:
The aim of the study is to investigate the correlation between the assumption of systemic medications (such as SSRI, PPI, anti-inflammatory drugs and anti-hypertensive drugs) and the failure of dental implant therapy in terms of occurrence peri-implantitis and/or implant failure.

The clinical records of all subjects treated with dental implants during the period between January 1st, 2005, and December 31st, 2020 in the Dental Clinic of the IRCCS Istituto Ortopedico Galeazzi (Milan, Italy) will be screened for inclusion.

Inclusion criteria: i) subjects who were 18 years old or older at the time of intervention; ii) subjects who provided their informed consent for the intervention iii) patients with total or partial edentulism treated with dental implants; iv) patients with at least 6 months follow-up, beginning from the date of placement of the prosthesis.

Exclusion criteria: i) incomplete data (e.g. absence of periapical radiographs) Descriptive statistics will be provided by means of mean values and standard deviations. Correlation between baseline parameters and outcomes will be provided through logistic regression. Survival tables and Kaplan-Meier analysis will be elaborated for survival analysis, considering the occurrence of implant failure and the diagnosis of peri-implantitis as events. Cox regression analysis will be used in order to evaluate the influence of the use of each drug on survival curves.

The level of significance was set at p<0.05. The sample size was calculated in order to evaluate the hazard risk of patients exposed to each specific drug (SSRI, PPI, Anti-inflammatory drugs or anti-hypertensive) compared to non-exposed patients. The ratio of exposed/non-exposed patients is expected to be 1:4 in the cohort. On the basis of a hypothesized 5-year incidence of peri-implantitis of 0.16, HR = 2, and a 10% dropout rate, the sample should be made of 358 subjects (72 exposed + 286 not exposed).

DETAILED DESCRIPTION:
Global demographic trends clearly show the increase in life expectancy and, as a direct consequence of progressive aging, the prevalence of disabling diseases with the relative intake of drugs. The intake of drugs such as thiazide diuretics, beta-blockers, anti-inflammatories, proton pump inhibitors and serotonin re-uptake inhibitors has been shown to be able to modulate bone metabolism with different mechanisms. Thus, they may be able to influence peri-implant health.

Proton pump blockers (PPIs) are a class of gastric acid secretion inhibitors that are currently among the best-selling drugs worldwide. The use of PPIs, especially at high doses and/or in long-term treatments, has been associated to an increased risk of hip, wrist and spine fractures. Different mechanisms have been suggested to explain the effects of PPIs on bone metabolism, which include: reduction of calcium absorption due to an increased pH in the small intestine; reduction of the osteoclastic resorption activity due to the modulation of vacuolar ATPase (V-ATPase) at the membrane level in the vesicles of osteoclasts; inhibition of non-specific alkaline phosphatase (ALP) and FOSFO1 in the vesicles of the bone matrix, increasing the expression of osteocalcin and the osteoprotegerin/RANKL ratio.

Selective serotonin reuptake inhibitors (SSRIs) are currently among the most common antidepressants and their main indications are major depression, generalized anxiety disorder, post-traumatic stress disorder, obsessive compulsive disorder, panic attack syndrome and bulimia. The action of selective serotonin reuptake inhibitors (SSRIs) on certain receptors and transporters such as 5-HT1B, 5-HT2B or 5-HT2C can result in impaired bone metabolism through increased differentiation and activation of osteoclasts. Reductions in bone mineral density (BMD) have been described, among others, in patients suffering from depressive syndromes which appear to be related to alterations in serotonin function. These findings suggest the hypothesis that SSRIs may have an impact also on the osseointegration process.

Anti-hypertensive drugs medications have been proven to interfere with bone metabolism through different mechanisms. For example, beta-blockers and angiotensin-converting enzyme inhibitors are able to inhibit osteoclasts activity by blocking the surface β-2 adrenergic receptors, which affects the renin-angiotensin system, while thiazides may enhance bone formation by increasing calcium absorption at the distal convoluted tubule.

Systemic corticosteroids are associated to various adverse reactions, especially when used at high doses or for long periods. Fracture and osteoporosis are among the most common corticosteroid-related adverse events.

The mechanism through which NSAIDs may negatively affect bone healing has not been fully explained, but it seems to be mostly related to the COX-2 blockade. Actually, it was proven that COX-2 is necessary for mesenchymal cells to differentiate into osteoblasts during fracture healing, while cele-coxib and other COX-2 blockers were reported to have a negative effect on the healing process by limiting osteogenesis and decreasing the osteogenic potential of mesenchymal stem cells.

The main aim of the study is to investigate if the systemic assumption of medications (such as SSRIs, PPIs, anti-inflammatory drugs, and anti-hypertensive drugs) could imply an increased risk of developing peri-implantitis.

Secondary aims will be to evaluate:

* the augmented risk of implant failure correlated to the assumption of drugs
* the correlation between the use of drugs and implant cumulative survival rate (CSR%)
* the relationship between drug dosage and the development of peri-implantitis
* relationship between drug dosage and implant failure The present will be a single-center, retrospective, observational, comparative study.

The definition of implant survival will be based on the fact that the implant is still in situ, stable, and supporting a functional prosthesis. An implant that was removed or spontaneously lost due to failed osseointegration will be considered an implant failure. Peri-implantitis will be defined according to the following parameters: 1) presence of bleeding and/or suppuration on gentle probing; 2) presence of radiographic bone loss of at least 2 mm, beyond crestal bone level changes due to initial bone remodeling, evaluated through comparison of baseline (one year after surgical intervention) and follow-up periapical radiographs; in absence of baseline periapical radiographs, presence of bone level located ≥ 3 mm apical to the most coronal portion of the intraosseous portion of the implant; 3) presence of an increased probing depth as compared to previous observations.

The following parameters will be collected from clinical records:

* Patient's age and sex at the time of surgical intervention
* description of systemic diseases (if any) at the time of surgical intervention
* description of pharmacological therapy (if any) at the time of surgical intervention
* smoking status (number of cigarettes (if reported)) at the time of surgical intervention
* history of periodontal disease before the surgical intervention or at the time of surgical intervention
* date of surgery
* implant position
* implant brand and type, diameter, length, diameter of the prosthetic platform
* characteristics of the bone regeneration procedure (if performed)
* description of surgical complications (if any)
* characteristics and timing of prosthetic rehabilitation (provisional and definitive)
* date of the last clinical control
* date of the last radiographic control
* failure occurrence date (if any)
* peri-implantitis occurrence date (if any)
* oral hygiene level
* frequency of maintenance recall sessions

Data collection will be performed in a maximum period of 5 months. Data analysis will take a maximum of 4 months, for a total duration of 9 months. The collected data refer to clinical records of patients treated with implants from January 1st, 2005 to June 30th, 2020 (last follow-up included: 6 month visit on December 2020).

The sample size was calculated in order to evaluate the hazard risk of patients exposed to a specific drug (SSRI, PPI, Anti-inflammatory drugs or anti-hypertensive) compared to non-exposed patients. The ratio of exposed/non-exposed patients is expected to be 1:4 in the cohort. The 5-year incidence in non-exposed patients in a previous series of cases resulted 0.16, and an HR=2 is expected in the exposed patients. On the basis of these assumptions, considering a 10% dropout rate, the sample should be made of 358 subjects (72 exposed + 286 not exposed ).

Therefore, a total of 358 patients who was exposed at least to one of the study drugs will be included: each subject will be evaluated both in the test group of the exposure drug (vs the group of subjects who did not take that drug), and in the control group for the drugs that he/she has not taken.

The calculation was performed using the method proposed by Schoenfeld. Descriptive statistics will be provided by means of mean values and standard deviations. Correlation between baseline parameters and outcomes will be provided through the use of logistic regression. Survival tables and Kaplan-Meier analysis will be elaborated for survival analysis, considering the occurrence of implant failure and the diagnosis of peri-implantitis as events. Cox regression analysis will be used in order to evaluate the influence of the use of SSRI and/or PPI on survival curves.

For all the analysis, the level of significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* subjects who were 18 years old or older at the time of intervention
* subjects who provided their informed consent for the intervention
* patients with total or partial edentulism treated with dental implants
* patients with at least 6 months follow-up, beginning from the date of placement of the prosthesis.

Exclusion Criteria:

* Incomplete data (e.g. absence of periapical radiographs)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The clinical records of all subjects treated with implants during the period between January 1st, 2005, and June 30th, 2020 in the Dental Clinic of the IRCCS Istituto Ortopedico Galeazzi (Milan, Italy) will be screened for inclusion
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Risk of peri-implantitis | 0 to 15 years
  Hazard risk of incurring in peri-implantitis in subjects assuming systemic medications (SSRIs, PPIs, anti-inflammatory drugs, and anti-hypertensive drugs)

SECONDARY OUTCOMES:
Influence of drugs on implant survival curves and peri-implantitis | 0 to 15 years
  Estimation of how the assumption of systemic medications could influence survival curves and the occurrence of peri-implantitis
Dosage and peri-implantitis | 0 to 15 years
  To establish if a relationship exists between the dosage of systemic medications and the risk of incurring in peri-implantitis
Dosage and implant failure | 0 to 15 years
  To establish if a relationship exists between the dosage of systemic medications and the risk of incurring in implant failure

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mombelli A, Cionca N. Systemic diseases affecting osseointegration therapy. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:97-103. doi: 10.1111/j.1600-0501.2006.01354.x. PMID 16968386
- [Background] Donos N, Calciolari E. Dental implants in patients affected by systemic diseases. Br Dent J. 2014 Oct;217(8):425-30. doi: 10.1038/sj.bdj.2014.911. PMID 25342349
- [Background] Vestergaard P. Skeletal effects of central nervous system active drugs: anxiolytics, sedatives, antidepressants, lithium and neuroleptics. Curr Drug Saf. 2008 Sep;3(3):185-9. doi: 10.2174/157488608785699432. PMID 18690999
- [Background] Brater DC. Update in diuretic therapy: clinical pharmacology. Semin Nephrol. 2011 Nov;31(6):483-94. doi: 10.1016/j.semnephrol.2011.09.003. PMID 22099505
- [Background] Gasiorowska A, Fass R. The proton pump inhibitor (PPI) test in GERD: does it still have a role? J Clin Gastroenterol. 2008 Sep;42(8):867-74. doi: 10.1097/MCG.0b013e31816c47ed. PMID 18645525
- [Background] Ye X, Liu H, Wu C, Qin Y, Zang J, Gao Q, Zhang X, He J. Proton pump inhibitors therapy and risk of hip fracture: a systematic review and meta-analysis. Eur J Gastroenterol Hepatol. 2011 Sep;23(9):794-800. doi: 10.1097/MEG.0b013e328348a56a. PMID 21701389
- [Background] Yu EW, Blackwell T, Ensrud KE, Hillier TA, Lane NE, Orwoll E, Bauer DC. Acid-suppressive medications and risk of bone loss and fracture in older adults. Calcif Tissue Int. 2008 Oct;83(4):251-9. doi: 10.1007/s00223-008-9170-1. Epub 2008 Sep 24. PMID 18813868
- [Background] Mattsson JP, Vaananen K, Wallmark B, Lorentzon P. Omeprazole and bafilomycin, two proton pump inhibitors: differentiation of their effects on gastric, kidney and bone H(+)-translocating ATPases. Biochim Biophys Acta. 1991 Jun 18;1065(2):261-8. doi: 10.1016/0005-2736(91)90238-4. PMID 1647821
- [Background] Roberts S, Narisawa S, Harmey D, Millan JL, Farquharson C. Functional involvement of PHOSPHO1 in matrix vesicle-mediated skeletal mineralization. J Bone Miner Res. 2007 Apr;22(4):617-27. doi: 10.1359/jbmr.070108. PMID 17227223
- [Background] Delomenede M, Buchet R, Mebarek S. Lansoprazole is an uncompetitive inhibitor of tissue-nonspecific alkaline phosphatase. Acta Biochim Pol. 2009;56(2):301-5. Epub 2009 Jun 18. PMID 19543559
- [Background] Mizunashi K, Furukawa Y, Katano K, Abe K. Effect of omeprazole, an inhibitor of H+,K(+)-ATPase, on bone resorption in humans. Calcif Tissue Int. 1993 Jul;53(1):21-5. doi: 10.1007/BF01352010. PMID 8102318
- [Background] Costa-Rodrigues J, Reis S, Teixeira S, Lopes S, Fernandes MH. Dose-dependent inhibitory effects of proton pump inhibitors on human osteoclastic and osteoblastic cell activity. FEBS J. 2013 Oct;280(20):5052-64. doi: 10.1111/febs.12478. Epub 2013 Sep 5. PMID 23937530
- [Background] Rodan GA, Martin TJ. Therapeutic approaches to bone diseases. Science. 2000 Sep 1;289(5484):1508-14. doi: 10.1126/science.289.5484.1508. PMID 10968781
- [Background] Haney EM, Warden SJ. Skeletal effects of serotonin (5-hydroxytryptamine) transporter inhibition: evidence from clinical studies. J Musculoskelet Neuronal Interact. 2008 Apr-Jun;8(2):133-45. PMID 18622082
- [Background] Schweiger U, Weber B, Deuschle M, Heuser I. Lumbar bone mineral density in patients with major depression: evidence of increased bone loss at follow-up. Am J Psychiatry. 2000 Jan;157(1):118-20. doi: 10.1176/ajp.157.1.118. PMID 10618024
- [Background] Rice JB, White AG, Scarpati LM, Wan G, Nelson WW. Long-term Systemic Corticosteroid Exposure: A Systematic Literature Review. Clin Ther. 2017 Nov;39(11):2216-2229. doi: 10.1016/j.clinthera.2017.09.011. Epub 2017 Oct 19. PMID 29055500
- [Background] Lisowska B, Kosson D, Domaracka K. Positives and negatives of nonsteroidal anti-inflammatory drugs in bone healing: the effects of these drugs on bone repair. Drug Des Devel Ther. 2018 Jun 21;12:1809-1814. doi: 10.2147/DDDT.S164565. eCollection 2018. PMID 29950815
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290